CLINICAL TRIAL: NCT04712279
Title: High-Dose Ivermectin for Mild-to-Moderate COVID-19 - The (HD)IVACOV Trial
Brief Title: The (HD)IVACOV Trial (The High-Dose IVermectin Against COVID-19 Trial)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corpometria Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORPO-DRUG-SARSCoV2-001
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: COVID-19; SARS-CoV-2; Covid19; Ivermectin
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ivermectin 0.6mg/kg/day (Active Comparator)
  Interventions: Drug: Ivermectin 0.6mg/kg/day; Drug: Hydroxychloroquine
- Ivermectin 1.0mg/kg/day (Active Comparator)
  Interventions: Drug: Ivermectin 1.0mg/kg/day; Drug: Hydroxychloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Ivermectin 0.6mg/kg/day — Use of ivermectin 0.6m/kg/day q.d.for 05 days
  Arms: Ivermectin 0.6mg/kg/day
Drug: Ivermectin 1.0mg/kg/day — Ivermectin 1.0mg/kg/day q.d. for 05 days
  Arms: Ivermectin 1.0mg/kg/day
Drug: Placebo — Placebo q.d.for 05 days
  Arms: Placebo
Drug: Hydroxychloroquine — Hydroxychloroquine 200mg/day q.d. for 05 days

SUMMARY:
Ivermectin, a classical antiparasitic and anti-scabies agent, has demonstrated antiviral activity for a variety of viruses including chikungunya virus, zyka virus and dengue virus and was tested as a potentially effective for COVID-19.

Although ivermectin demonstrated potent in vitro action by reducing viral load by 5000x after 48 hours of incubation, simultaneous pharmacokinetics simulations suggested that the minimum effective concentrations would be unfeasible to be reached within safety range (EC-50 = 2 Micromol).

However, despite the theoretical unfeasible concentrations to be achieved, preliminary observational yet well-structured studies followed by randomized clinical trials (RCTs) demonstrated ivermectin efficacy when combined with hydroxychloroquine, doxycycline or azithromycin, which was corroborated by a recent systematic review and metanalysis. In common, a dose-response effect for effectiveness was observed, and no adverse effects was reported at any dose between 0.2mg/kg/day and 1.0mg/kg/day.

Based on the scientific rationale combined with the preliminary evidence, ivermectin has sufficient evidence to be tested in higher doses in a RCT for COVID-19. The investigators propose to test ivermectin at high doses as a treatment for patients recently diagnosed with COVID-19, aiming to explore the possible protective role of high-dose ivermectin in SARS-CoV-2 infection in terms of reduction of clinic and virologic disease duration, and prevention of oxygen use, hospitalization, mechanical ventilation, death, and post-COVID persisting symptoms.

DETAILED DESCRIPTION:
Overall

COVID-19 is a multisystemic disease caused by SARS-CoV-2 that has become a pandemic largely due to a combination of favorable transmission and infection characteristics for its spread, including prolonged preclinical or also asymptomatic yet transmitting period, relatively highly resistant to mechanical and physical barriers and prolonged survival in the air, and transmission patterns not yet fully elucidated.

While vaccines are not widely available, the number of new cases should not decrease dramatically, unfortunately, since a large percentage of the population has not been infected by the SARS-CoV-2 yet, reinfection becomes increasingly plausible with mutations in the virus, and virus contention policies failed to be 100% effective.

Considering potential antiviral approaches for COVID-19, their effectiveness only make sense if tested and given early in the disease, during viral dissemination. The learning that oseltamivir is only effective for Influenza A in the first three days of disease finds strong plausibility, and reinforces the expected lack of effectiveness of any drug with in vitro or preliminary antiviral activity reported when tested in hospitalized or non-mild patients, once COVID-19 presents tend to present mild symptoms during the viral dissemination stage.

An actual early detection of COVID-19, i.e., before its progression to further inflammatory stages, is challenging, once the earliest symptoms tend to be unspecific, mild, and hardly attributable to COVID-19. By suspecting of COVID-19 in the presence of any symptom, specific to COVID-19 or not, sensitivity was met to be above 90% while specificity was also relatively high (above 50%). In addition, time-to-treat, rather than which drug to choose, could better determine the effectiveness of a specific approach.

Ivermectin: potential antiviral activity for COVID-19

Among drugs potentially effective for COVID-19, despite the classical antiparasitic and anti-scabies use, ivermectin has demonstrated antiviral activity for a variety of viruses by inhibiting and reducing the viral shedding duration, including chikungunya and other alphaviruses, zyka virus, dengue virus and other simple-strain RNA viruses.

In the search for drugs with anti-SARS-CoV-2 activity, considering its effects on other viruses, ivermectin was tested in a Vero-hSLAM cell model and demonstrated potent in vitro action, by reducing viral load by 5000x after 48 hours of incubation. However, after initial promising results, simultaneous pharmacokinetics simulations suggested that the minimum effective concentrations would be unfeasible to be reached within safety range (EC-50 = 2 Micromol).

Although the theoretical minimum concentration required for antiviral action was apparently at least 17 times higher than the lethal dose and up to 10,000 times the usually prescribed doses for humans ( IC50 of 2.2 - 2.8 µM for monkeys), which would reduce the chances of ivermectin efficacy for COVID-19, preliminary observational yet well-structured studies demonstrated substantial synergistic action of ivermectin when added to "standard of care", usually hydroxychloroquine with or without macrolides. In a specific study, the use of ivermectin, even in low doses, reduced by 40% the absolute risk of death among patients more severely affected by COVID-19.

Some randomized clinical trials (RCTs) demonstrated efficacy of ivermectin when combined with hydroxychloroquine, doxycycline or azithromycin, in both mildly (and presumedly early) and more severely affected subjects with COVID-19. Demonstrated benefits included lower disease progression and reduced COVID-related mortality.

In comparative analyses, combinations between ivermectin and azithromycin, doxycycline or hydroxychloroquine demonstrated superiority compared to combinations between hydroxychloroquine and azithromycin or hydroxychloroquine alone.

The exact mechanisms of action remain nuclear. At least one study employing higher doses (0.6mg/kg/day) demonstrated in vivo antiviral activity, but only when maximum concentration reached serum levels above 160 ng/ml, which only occurred in 45% of subjects, even at higher doses. The antiviral mechanisms include modification in the ACE-2 glycation patterns, inhibition of the viral Helicase (NSP13) and disruption of the alpha-importin heterodimer.

In a recent systematic review and metanalysis, a dose-response correlation has also been observed in terms of endpoints, reinforcing the role of ivermectin as actins as an anti-SARS-CoV-2 action drug. However, even in lower doses ivermectin was able to demonstrate clinical benefits, allowing the hypothesis that ivermectin also exerts anti-inflammatory effects, which could include the blockage of STAT-1 migration to the nucleus, and could justify its use even at later stages of the disease.

Collectively, higher yet safe ivermectin doses find stronger plausibility and preliminary evidence to be tested in RCTs. In addition, approaches to increase ivermectin absorption and bioavailability should be encouraged.

Based on the scientific rationale combined with preliminary evidence, ivermectin has sufficient evidence to be tested at higher doses in a RCT for COVID-19. The investigators propose to test ivermectin at high doses as a treatment for patients recently diagnosed with COVID-19. This study is intended to explore the possible protective role of high-dose ivermectin in SARS-CoV-2 infection in terms of reduction of clinic and virologic disease duration, and prevention of oxygen use, hospitalization, mechanical ventilation, death, and post-COVID persisting symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory or clinically confirmed positive SARS-CoV-2 rtPCR test (AndroCoV Clinical Scoring for COVID-19 Diagnosis1) within 7 days prior to randomization
2. ≥18 years old
3. Laboratory confirmed positive SARS-CoV-2 rtPCR test within 7 days prior to randomization
4. Clinical status on the COVID-19 Ordinal Scale (defined in Section 5.1) of 1 to 3
5. Subject (or legally authorized representative) gives written informed consent prior to performing any study procedures
6. Subject (or legally authorized representative) agree that subject will not participate in another COVID-19 trial while participating in this study

Exclusion Criteria:

1. Subject enrolled in a study to investigate a treatment for COVID-19
2. Require oxygen use, hospitalization or mechanical ventilation
3. Tachycardia (HR > 150 bpm) or hypotension (BP < 90/60 mmHg)
4. Patients who are allergic to the investigational product or similar drugs (or any excipients);
5. Subjects with QTcF > 450 ms
6. Subjects with uncontrolled medical conditions that could compromise participation in the study - uncontrolled hypertension (BP > 220/120 mmHg), uncontrolled hypothyroidism (TSH > 10 iU/L), uncontrolled diabetes mellitus (HbA1c > 12%)
7. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
8. Estimated glomerular filtration rate (eGFR) < 30 ml/min or requiring dialysis
9. Subject (or legally authorized representative) not willing or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2021-03-21 (Estimated); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
World Health Organization (WHO) Clinical Progression Scale [0 to 10; 0 = uninfected; 10 = death] | Day 14
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by World Health Organization (WHO) Clinical Progression Scale [0 to 10; 0 = uninfected; 10 = death]

SECONDARY OUTCOMES:
World Health Organization (WHO) COVID=19 Ordinal Scale for Clinical Improvement [1 to 8; 1 = not hospitalized, no limitation on activities; 8 = death] [Time Frame: Day 7] | Day 7
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by World Health Organization (WHO) COVID=19 Ordinal Scale for Clinical Improvement [1 to 8; 1 = not hospitalized, no limitation on activities; 8 = death]
Time-to-recovery | Day 28
  Recovery is defined as the first day on which the subject satisfies category one from the COVID ordinal scale (defined in Section 5.1): (1) Not hospitalized, no limitations on activities. [Parameter: Number of days until achieve Category 1 of the World Health Organization (WHO) COVID=19 Ordinal Scale for Clinical Improvement [1 to 8; 1 = not hospitalized, no limitation on activities; 8 = death]
Viral load | Day 5
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by viral load measured by rtPCR-SARS-CoV-2 (CTs)
Positivity rate of rtPCR-SARS-CoV-2 (qualitative analysis) | Day 5
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by viral load measured by positivity rate (% of positive, detected rtSARS-CoV-2)
Duration of fatigue | Day 14
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by duration of fatigue (days)
Duration of anosmia | Day 14
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by duration of anosmia (days)
Overall duration of clinical manifestations | Day 14
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by duration of overall symptoms (days)
Proportion of subjects needing additional drugs or interventions | Day 28
  Defined as the number of subjects who have required additional drugs (glucocorticoids, anticoagulants, etc) or interventions allocated to each arm divided by the number of subjects randomized to that specific arm (%). Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the proportion of subjects needing additional drugs or interventions in each arm.
Proportion of subjects needing oxygen use | Day 28
  Defined as the number of subjects who have required oxygen use allocated to each arm divided by the number of subjects randomized to that specific arm (%). Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the proportion of subjects needing oxygen use in each arm.
Proportion of subjects needing high-flow oxygen therapy or non-invasive ventilation | Day 28
  Defined as the number of subjects who have required high-flow oxygen use or non-invasive mechanical ventilation allocated to each arm divided by the number of subjects randomized to that specific arm (%). Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the proportion of subjects needing high-flow oxygen use or non-invasive mechanical ventilation in each arm.
Proportion of hospitalizations | Day 28
  Defined as the number of hospitalizations in each arm divided by the number of subjects randomized to that specific arm (%). Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the proportion of hospitalizations in each arm.
Proportion of mechanical ventilation use | Day 28
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of mechanical ventilation use in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of pressors use | Day 28
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects needing use of pressors in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of deaths | Day 28
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects who have died in each arm divided by the numbers of subjects randomized to the treatment arm (%).
Proportion of post-COVID mental symptoms | Day 30
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects persisting with mental symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of post-COVID mental symptoms | Day 60
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects persisting with mental symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of post-COVID mental symptoms | Day 90
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects persisting with mental symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of post-COVID physical symptoms | Day 30
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects persisting with physical symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of post-COVID physical symptoms | Day 60
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects persisting with physical symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of post-COVID physical symptoms | Day 90
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects persisting with physical symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of post-COVID overall symptoms | Day 30
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects persisting with any symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of post-COVID overall symptoms | Day 60
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects persisting with any symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%).
Proportion of post-COVID overall symptoms | Day 90
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects persisting with any symptoms after COVID-19 resolution in each arm divided by the number of subjects randomized to that specific arm (%).
Duration of new oxygen use | Day 28
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the duration of new oxygen use measured in days among subjects that did not require oxygen upon randomization and required oxygen use after the beginning of treatment, in each arm (days)
Duration of hospitalization | Day 28
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the duration of hospitalization measured in days among subjects that required hospitalization, in each arm (days)
Duration of mechanical ventilation | Day 28
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the duration of mechanical ventilation measured in days among subjects that required mechanical ventilation, in each arm (days)
Proportion of increased ultrasensitive C-reactive protein (usCRP) (defined as usRCP > 7 mg/L) | Day 1
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting increased ultrasensitive C-reactive protein (usCRP) at Days 1, 2, 3 and 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of increased ultrasensitive C-reactive protein (usCRP) (defined as usRCP > 7 mg/L) | Day 3
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting increased ultrasensitive C-reactive protein (usCRP) at Days 1, 2, 3 and 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of increased ultrasensitive C-reactive protein (usCRP) (defined as usRCP > 7 mg/L) | Day 7
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting increased ultrasensitive C-reactive protein (usCRP) at Days 1, 2, 3 and 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of decrease in erythrocyte sedimentation rate (ESR) (defined as ESR decrease > 50% compared to Day 1) | Day 1
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting ESR decrease > 50% at Days 2, 3 and 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of decrease in erythrocyte sedimentation rate (ESR) (defined as ESR decrease > 50% compared to Day 1) | Day 3
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting ESR decrease > 50% at Days 2, 3 and 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of decrease in erythrocyte sedimentation rate (ESR) (defined as ESR decrease > 50% compared to Day 1) | Day 7
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting ESR decrease > 50% at Days 2, 3 and 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of increase in eosinophils (defined as eosinophils increase > 50% compared to Day 1) | Day 1
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting eosinophils increase > 50% at Days 2, 3 and 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of increase in eosinophils (defined as eosinophils increase > 50% compared to Day 1) | Day 3
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting eosinophils increase > 50% at Days 2, 3 and 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of increase in eosinophils (defined as eosinophils increase > 50% compared to Day 1) | Day 7
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting eosinophils increase > 50% at Days 2, 3 and 7, divided by the number of subjects randomized to that specific arm (%).
Proportion of increased d-dimer (defined as d-dimer > 500 mg/dL) | Day 7
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by the number of subjects presenting increased d-dimer protein (usCRP) at Day 7, divided by the number of subjects randomized to that specific arm (%).
Disease duration | Day 14
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by duration of symptoms, complications, or any other COVID-related clinical or biochemical sign of disease
Change in viral load from baseline to Day 5 | Day 30
  Treatment efficacy of high-dose Ivermectin relative to placebo arm as assessed by change in viral load from baseline to Day 5 measured by rtPCR-SARS-CoV-2 (CTs)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Zimerman, MD, Study Director — Corpometria Institute; Flavio A Cadegiani, MD, PhD, Principal Investigator — Corpometria Institute; Applied Biology

REFERENCES:
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Result] Li L, Liu J, Qin K. Comparison of double-dose vs standard-dose oseltamivir in the treatment of influenza: A systematic review and meta-analysis. J Clin Pharm Ther. 2020 Oct;45(5):918-926. doi: 10.1111/jcpt.13203. Epub 2020 Jun 4. PMID 32497319
- [Result] Varghese FS, Kaukinen P, Glasker S, Bespalov M, Hanski L, Wennerberg K, Kummerer BM, Ahola T. Discovery of berberine, abamectin and ivermectin as antivirals against chikungunya and other alphaviruses. Antiviral Res. 2016 Feb;126:117-24. doi: 10.1016/j.antiviral.2015.12.012. Epub 2016 Jan 2. PMID 26752081
- [Result] Padhy BM, Mohanty RR, Das S, Meher BR. Therapeutic potential of ivermectin as add on treatment in COVID 19: A systematic review and meta-analysis. J Pharm Pharm Sci. 2020;23:462-469. doi: 10.18433/jpps31457. PMID 33227231
- [Result] Rajter JC, Sherman MS, Fatteh N, Vogel F, Sacks J, Rajter JJ. Use of Ivermectin Is Associated With Lower Mortality in Hospitalized Patients With Coronavirus Disease 2019: The Ivermectin in COVID Nineteen Study. Chest. 2021 Jan;159(1):85-92. doi: 10.1016/j.chest.2020.10.009. Epub 2020 Oct 13. PMID 33065103
- [Result] Elgazzar, A et al. Efficacy and Safety of Ivermectin for Treatment and prophylaxis of COVID-19 Pandemic. Research Square doi.org/10.21203, 2020
- [Result] Chowdhury, ATMM et al. A Randomized Trial of Ivermectin-Doxycycline and Hydroxychloroquine-Azithromycin therapy on COVID19 patients. Research Square: https://doi.org/10.21203/rs.3.rs-38896/v1, 2020.
- [Result] Niaee, MS et al. Ivermectin as an adjunct treatment for hospitalized adult COVID-19 patients: A randomized multi-center clinical trial. Research Square: https://doi.org/10.21203/rs.3.rs-109670/v1, 2020.
- [Result] Francés-Monerris, A et al. Has Ivermectin Virus-Directed Effects against SARS-CoV-2? Rationalizing the Action of a Potential Multitarget Antiviral Agent. ChemRxiv, 2020.